CLINICAL TRIAL: NCT04014634
Title: GON-injection for a Sooner and Better Treatment of Cluster Headache: a Double-blind Randomized Controlled Trial
Brief Title: GON-injection for a Sooner and Better Treatment of Cluster Headache
Acronym: CHIANTI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Netherlands Brain Foundation (Other); Innovatiefonds Zorgverzekeraars (Other)
Responsible Party: Principal Investigator, RolfFronczek, Principal investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL6719705818
Record Dates: First submitted 2019-07-08; First posted 2019-07-10 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Cluster Headache, Episodic; Greater Occipital Nerve Injection
MeSH Terms: conditions — Cluster Headache | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Injection of NaCl
  Interventions: Other: Placebo
- Verum (Experimental)
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — Single GON injection with methylprednisolone
  Arms: Verum
Other: Placebo — Single GON-injection with NaCl
  Arms: Placebo

SUMMARY:
Cluster headache is a very severe primary headache disorder. In episodic cluster headache, attacks occur in 'bouts' (clusters) lasting weeks to months. Management of cluster headache entails a combination of attack and prophylactic treatment. Current first choice prophylactic treatment (verapamil) has considerable side effects which can be serious and include possibly fatal cardiac arrhythmias; and it can take weeks to titrate to an effective dose. Evidence has emerged that local steroid injection of the greater occipital nerve (GON) may be effective in cluster headache, but this method has not been investigated as a first line prophylactic treatment in a large, well-documented group of episodic cluster headache patients who are still free of prophylactic medication and just entered a new cluster headache episode. As such, GON-injection has not yet found its way into current treatment protocols. The investigators plan to perform this multicentre double-blind randomized controlled trial to investigate whether GON-injection is efficacious as a first-line prophylactic treatment, aiming to remove the need for high doses of daily medication - such as verapamil - with associated side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to be diagnosed with episodic cluster headache according to the international classification of headache disorders - third edition, ICHD-3
* Patients have to be aged 18-65 years
* Patients need to be newly diagnosed and treatment naïve, or already diagnosed and currently free from prophylactic treatment
* Patients need to have a mean of 1 or more attacks per day in the 3 days preceding inclusion.
* Patients should be in their cluster period for shorter than 4 weeks before inclusion.

Exclusion Criteria:

* A contraindication for treatment with steroids or verapamil
* The use of anticoagulants or known bleeding disorder.
* Use of any prophylactic medication for cluster headache
* Patients with a history of other primary headache who are currently using prophylactic medication for this headache
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Verapamil mean total dose | 12 week period
  Difference in mean total dose of verapamil used during the study period

SECONDARY OUTCOMES:
Days to remission | 12 weeks
  Median number of days to remission (7 consecutive days without attack)
Daily attacks | 12 weeks
  Mean number of attacks per day during the study period
Peak dose verapamil | 12 weeks
  Peak dose verapamil
Preamature termination | 12 weeks
  Premature termination of study due to need for escape medication

OTHER OUTCOMES:
Use of attack medication | 12 weeks
  The total use of attack medication (stratified for oxygen and sumatriptan)
Daily attack severity and duration | For the total study period and each of the three consecutive 4-week time periods
  Mean number, severity (1-10) and duration of attack per day.
Attack-freedom | days 7, 14 and 28
  Percentage of patients that are attack-free at days 7, 14 and 28
Non-cluster headache | 12 weeks
  Occurrence of 'non-cluster' headache (number of days and mean intensity per affected day)
Adverse events | 12 weeks
  Percentage of subjects with adverse-events (stratified for type of side effect (AE, SAE, SUSAR))
Subjective feeling | Days 7, 14 and 28
  Subjective feeling at days 7, 14 and 28 (visual analogue scale, VAS. Scale from 0 to 10 where 0 is worst imaginable and 10 best imaginable)
Satisfaction score | 12 weeks
  Satisfaction score (7 point scale, 0 to 6. 0 is completely unsatisfied and 6 completely satisfied)
Recommendation | Days 7, 14 and 28
  Would the patient recommend this treatment to others
Blinding participants | Days 7, 14 and 28
  What treatment does the patient think he/she received (placebo/GON/uncertain)
Blinding investigators | Days 7, 14 and 28
  What treatment do the investigators think the patient has had

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Fronczek, MD, PhD, Principal Investigator — LUMC
Locations (6):
- Netherlands (6):
  - Boerhaave Clinics, Amsterdam, North Holland
  - LUMC, Leiden, South Holland
  - Alrijne Ziekenhuis, Leiderdorp, South Holland
  - Tergooi Ziekenhuis, Blaricum
  - Zuyderland Medisch Centrum, Heerlen
  - Canisius-Wilhelmina Hospital, Nijmegen

IPD SHARING:
Plan to Share IPD: No
All Data will be stored using Castor EDC. All hard copies will be stored in the individual centers. If requested, after study completion, data can be shared with de PIs in participating centers.

REFERENCES:
- [Derived] Brandt RB, Mulleners WM, Couturier E, Carpay JA, Gerlach OHH, Niesters M, Haan J, van Zwet EW, Ferrari MD, Fronczek R. Greater occipital nerve injection with methylprednisolone as transitional therapy in episodic cluster headache: Results from an RCT. Cephalalgia. 2025 Sep;45(9):3331024251370324. doi: 10.1177/03331024251370324. Epub 2025 Sep 24. PMID 40990636